CLINICAL TRIAL: NCT01796275
Title: A "Happy Family Kitchen" Initiative for Promoting Family Health, Happiness, and Harmony in Tsuen Wan, Kwai Chung and Tsing Yi District
Brief Title: Happy Family Kitchen Project II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Council of Social Service (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HFK2
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Family Communication; Family Health; Happiness and Harmony

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Subjects will have a core session intervention and booster intervention; questionnaire evaluation is conducted at baseline, post-session, pre-booster and 3 month after core session.
  Interventions: Behavioral: Core intervention program; Behavioral: Booster session
- Group B (Experimental): Subjects will only have a core session intervention; Questionnaire evaluation are conducted at baseline (T1-baseline), post-session (T2), 4 weeks after core session (T3) and 3 month after core session (T4).
  Interventions: Behavioral: Core intervention program
- Group C (Other): Group C is a waiting list control, only questionnaire evaluations can be conducted at T1-baseline, T3- tea gathering and T4- 3 month after baseline evaluation; when finish T4 evaluation, the core session and booster can be optionally conducted subsequently.
  Interventions: Behavioral: Control only (Tea gathering)

INTERVENTIONS:
Behavioral: Core intervention program
  Arms: Group A; Group B
Behavioral: Booster session
  Arms: Group A
Behavioral: Control only (Tea gathering)
  Arms: Group C

SUMMARY:
The School of Public Health of HKU collaborates with the Hong Kong Council of Social Service (HKSCC) to conduct a district-based mega-project "Happy Family Kitchen", which using "eating" and "the kitchen" as a platform, to make the effort to improve effective communication in Hong Kong families.

The "HFK 2" project is a enhanced version of HFK project, which plan to be conducted in the Tsuen Wan, Kwai Chung and Tsing Yi district from August 2012 to August 2013. This project adopts a cluster-randomized controlled design, with the application of positive psychology concepts as a theoretical framework. A community-based participatory (CBP) approach, which is an effective way to engage public health researchers and community members (NGOs, schools, other major stakeholders, and participants), will be used. Both quantitative and qualitative methods will be used in the evaluation of major outcomes (participants' family relationship and 3Hs) at different time points throughout the project. Process evaluation will be performed to evaluate the process of each component of the project. The whole project includes two phases:

Phase 1: Model enhancement- an enhanced model of project is started with the training the trainer workshop to build capacity among the community partners. After that, the trained community partners design and conduct the district-based intervention programmes by using one of the five themes of the positive psychology framework, which teach the participants to practice positive behaviors for improving family communication, and in turn promote the 3Hs. The five themes are joy, flow, gratitude, savoring and listening. The pre-, post-, 4 weeks and 3 month follow up questionnaire surveys are conducted to assess the effectiveness of the programmes. All of the participating NGOs and schools will be randomly allocated into three groups:

Intervention arm 1: core session intervention + booster intervention; Intervention arm 2: only core session intervention; Control arm: waiting list control, only questionnaire evaluations can be conducted at different time points.

A subsequent qualitative study is conducted to further explore the outcomes, the problems and the requirements from the programmes.

Phase 2: Model scaling up- A series of Professional Tool Kits consist of practice guides and evaluation tools for different service settings will be published with the contribution of participating NGOs and project partners. The tool kits will be the key reference and be further disseminated to a wider scope. A series of Professional Practice Seminars will be organized in different regions (including Hong Kong, Kowloon and New Territories). Social work practitioners of various service settings will be invited to attend the seminars. The evidence-based professional tool kits will be introduced and distributed in the seminar. Clinical psychologist will be the speaker on how to apply positive psychology in practice, and HKU staff will also illustrate the use of evaluation tools in assessing the outcome of the program. Participating NGOs of this project will be invited to share their practice experience in Tsuen Wan and Kwai Tsing district as well. another new edition of Happy Family Cookbook will be published and distributed to the whole territory. The new edition will be enhanced with more attractive content including healthy recipes and tips for positive communication etc. To enhance the interactivity of the cookbook, related apps for mobile devices will be developed for public free download.

DETAILED DESCRIPTION:
Background

Traditionally, Chinese people place great importance on their families. However, the increasingly busy city lifestyle leaves little time for family gatherings and communication. A recent census by the Hong Kong government showed that nearly 50% of respondents never, or only occasionally, listened to their parents' concerns or heeded their advice on important matters; and over 50% rarely or never listened to their siblings' views or gave them advice on important matters. This lack of communication raises the problem of neglect or indifferent, rigid relationships within the family, which tend to exert negative effects on health, happiness and harmony (the 3Hs). For these reasons, the School of Public Health of HKU collaborates with the Hong Kong Council of Social Service (HKSCC) to conduct a district-based mega-project "Happy Family Kitchen", which using "eating" and "the kitchen" as a platform, to make the effort to improve effective communication in Hong Kong families.

Current evidence

The Happy Family Kitchen 1 project (HFK 1 project) was launched in September 2010 with the mission to promote family health, happiness and harmony (i.e. 3Hs) by advocating positive family communication. In collaboration with 18 NGOs and SWD (including 23 service units) in Yuen Long district, the one-year HFK project was completed in August 2011, with the following achievements:

* Over 1,000 families joined the 23 community programs under the project theme of positive family communication in Yuen Long district.
* 50 professional social work practitioners were equipped with knowledge and skills in integrating positive psychology and program design through trainer's training.
* Built-in evaluative research study conducted to examine the project process and outcome.
* Practice wisdom consolidated and shared with the social services sector through a sharing forum and a specially designed practice manual.
* Over 10,000 pieces of Happy Family Kitchen Cookbook were distributed to the public with positive feedback received.
* Series of media publicity (e.g. news feature, magazine, Roadshow, You tube etc) was conducted to convey the key message of promoting positive family communication.

Upon completion of the one-year pilot project, it was observed that substantial impact was made in various aspects, namely:

i. Participating Families - over 1,000 families in Yuen Long district participated in the community programs and learned the ways to enhance the communication with their family members through the means of dinning together.

ii. Social Work Practice - prototype of the practice model adopting positive psychology (i.e. 正向溝通五常法) was successfully piloted with empirical evidence supported. Practice wisdom of applying such model had been documented as practice manual for future use. Besides, evidence-based practice approach was promoted by supporting NGOs to integrate theoretical framework (i.e. positive psychology) and program evaluation into practice.

iii. Community Partnership - district-based collaboration network among NGOs and SWD established for joint effort in promoting 3Hs in the community. Family-centered approach had been adopted as the foundation of collaboration among service units of different settings.

iv. Territory-wide Public Education - the key message on encouraging positive family communication was disseminated to the whole territory through series of publicity work. The impact of the project was beyond Yuen Long district.

The community-based HFK project was the first of its kind which aimed to integrate the best social work practice with public health science. Based on the successful experience of the HKF project in Yuen Long district, it is crucial to think of ways to sustain the project impact in the longer term. As the enhanced version of the HFK project, HFK2 is going to answer this question by suggesting three possible ways forward:

i) enhancing the existing practice model with evidence support; ii) scaling up the practice model in wider scope; and iii) strengthening the key message of promoting positive family communication in the society.

Aim and objectives The aim of this study is to assess the effectiveness of a district-based intervention programme (with the application of positive psychology) among families in the Tsuen Wan, Kwai Chung and Tsing Yi district, on enhancing their family communication and family 3Hs.

The specific objectives of the study include:

i. To promote family happiness, harmony and health by building capacity for families on positive communication.

ii. To enhance and test the practice model integrating positive psychology and family education.

iii. To improve and strengthen the community-based service model and keep sustainable application in the target district

Hypotheses

Primary hypothesis:

Families participated in a district-based programme that received a positive psychology intervention (intervention groups) have better family communication and family 3Hs than families who don't participate in a community-based programme (control group) during 3 months.

Second hypotheses:

i. The district-based intervention programmes (core session) has significant effect on improving family communication and 3Hs (intervention 2 versus control) ii. The District-based intervention programmes (whole dosage, core session +booster) have significant effect on improving family communication and 3Hs (intervention 1 versus control) iii. Booster intervention can further improve the family communication and 3Hs compares with non-booster intervention (intervention 1 versus intervention 2)

Randomization

A total of 30 NGOs and schools will be randomized into three groups respectively:

Intervention arm 1: core session intervention + booster intervention; questionnaire evaluation is conducted at baseline (T1), post-session (T2), pre-booster (T3) and 3 month after core session (T4-tea gathering).

Intervention arm 2: only core session intervention; once finish the T4 evaluation, the booster can be conducted subsequently. Questionnaire evaluation are conducted at baseline (T1), post-session (T2), T3 and 3 month after core session (T4- tea gathering).

Control arm: waiting list control, only questionnaire evaluations can be conducted at T1(Tea gathering), T3(Tea gathering) and T4; when finish T4 evaluation, the core session and booster can be conducted subsequently.

ELIGIBILITY:
Inclusion criteria:

1. For the district-based programmes, and focus groups of participants:

   Participants aged six or above, who can communicate with social workers, and who are currently residing in Tsuen Wan, Kwai Chung and Tsing Yi District /are service users of the corresponding NGO/ are students in Tsuen Wan, Kwai Chung and Tsing Yi District. Participants who are between six and eight years old are required to be assisted individually by social workers in completing questionnaires.
2. For the social workers' training programme, the health education forum, the practice wisdom forum and focus groups of social workers:

   Social or community workers who can read Chinese and speak Cantonese, and are currently working in selected social service organizations or government agencies in the Tsuen Wan, Kwai Chung and Tsing Yi District.
3. In-depth interviews of community stakeholders: community stakeholders who can read Chinese and speak Cantonese, and are currently working in the social service organizations (participate or not participant in this project) or government agencies in the Tsuen Wan, Kwai Chung and Tsing Yi District.

Exclusion Criteria:

* Participants who fail to meet the inclusion criteria

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes in family communication from baseline to 3 months after intervention | Pre-intervention (Up to 2 days before), immediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Family communication will be assessed by the Family communication scale.
Changes in family happiness from baseline to 3 months after intervention | Pre-intervention (Up to 2 days before), immediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Happiness will be determinded by Subjective Happiness Scale and the one item question adopted from Subramanian et al. Self- preceived happiness at the individual and family level will aso be assessed by a 0-10 score at 4 time points.
Changes in family health from baseline to 3 months after intervention | Pre-intervention (Up to 2 days before), immediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Health will be evaluated by the SF-12v2 Health Survey. Harmony will be assessed by a 12-item scale. Self-preceived health, at the individual and family level will also be assessed by a 0-10 score at 4 time points.
Changes in family harmony from baseline to 3 months after intervention | Pre-intervention (Up to 2 days before), immediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Harmony will be assessed by a 12-item scale. Self-preceived harmony, at the individual and family level will also be assessed by a 0-10 score at 4 time points.

SECONDARY OUTCOMES:
Changes in Participants' attitudes towards performing the suggested behaviours from baseline to 3 months after intervention | Pre-intervention (Up to 2 days before), immediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Questionnaire will be used to evaluate the changes in participants' attitude towards performing the suggested behaviors from baseline to 3 months after intervention.
Changes in Participants' intention at performing the suggested behaviours from baseline to 3 months after intervention | Pre-intervention (Up to 2 days before), immediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Questionnaire will be used to evaluate the changes in participants' intention at performing the suggested behaviors from baseline to 3 months after intervention.
Changes in Participants' frequency of performing the suggested behaviours from baseline to 3 months after intervention | Pre-intervention (Up to 2 days before), immediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Questionnaire will be used to evaluate the changes in participants' frequency of performing the suggested behaviors from baseline to 3 months after intervention.
Changes in social workers' knowledge of the application of positive psychology in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' knowledge of the application of positive psychology in the CBPR project before and after the training session.
Changes in social workers' attitudes of the application of positive psychology in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' attitudes of the application of positive psychology in the CBPR project before and after the training session.
Changes in social workers' self-competence of the application of positive psychology in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' self-competence of the application of positive psychology in the CBPR project before and after the training session.
Changes in social workers' knowledge of the application of logic model in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' knowledge of the application of logic model in the CBPR project before and after the training session.
Changes in social workers' attitudes of the application of logic model in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-upediate post- intervention (Up to 2 weeks after), four weeks and three months after intervention.
  Questionnaire will be used to investigate the changes in social workers' attitudes of the application of logic model in the CBPR project before and after the training session.
Changes in social workers' self-competence of the application of logic model in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' self-competence of the application of logic model in the CBPR project before and after the training session.
Changes in social workers' knowledge of the application of process evaluation in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' knowledge of the application of process evaluation in the CBPR project before and after the training session.
Changes in social workers' attitudes of the application of process evaluation in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' attitudes of the application of process evaluation in the CBPR project before and after the training session.
Changes in social workers' self-competence of the application of process evaluation in the CBPR project before and after training session | Pre- and post- training (Up to 2 weeks before and after) ; as well as a 6-month, and 12-month follow-up
  Questionnaire will be used to investigate the changes in social workers' self-competence of the application of process evaluation in the CBPR project before and after the training session.
The social impact of the CBPR project | Post intervention program (Up to 3 months after)
  Evaluated by conducting community stakeholders' in-depth interviews.
The process of community based intervention programme | Observe in every session of the community based intervention programme, including core intervention sessions, booster sessions, and tea-gathering sessions.
  Assessed by a Process Evaluation on-site observation form, and a series of checklists including Resources input record sheet, Participants' attendance form, Programme rundown, Attendance record form, and NGOs' final report. The components of process evaluation, including context, reach, dose delivered, dose received, fidelity and recruitment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia SC Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Council of Social Service, Hong Kong, China

REFERENCES:
- [Derived] Lai AY, Stewart SM, Mui MW, Wan A, Yew C, Lam TH, Chan SS. An Evaluation of a Train-the-Trainer Workshop for Social Service Workers to Develop Community-Based Family Interventions. Front Public Health. 2017 Jun 30;5:141. doi: 10.3389/fpubh.2017.00141. eCollection 2017. PMID 28713801
- [Derived] Ramirez-Velez R, Tordecilla-Sanders A, Tellez-T LA, Camelo-Prieto D, Hernandez-Quinonez PA, Correa-Bautista JE, Garcia-Hermoso A, Ramirez-Campillo R, Izquierdo M. Effect of Moderate- Versus High-Intensity Interval Exercise Training on Heart Rate Variability Parameters in Inactive Latin-American Adults: A Randomized Clinical Trial. J Strength Cond Res. 2020 Dec;34(12):3403-3415. doi: 10.1519/JSC.0000000000001833. PMID 28198783
- [Derived] Ho HC, Mui M, Wan A, Ng YL, Stewart SM, Yew C, Lam TH, Chan SS. Happy Family Kitchen II: a cluster randomized controlled trial of a community-based positive psychology family intervention for subjective happiness and health-related quality of life in Hong Kong. Trials. 2016 Jul 29;17:367. doi: 10.1186/s13063-016-1508-9. PMID 27473842
- [Derived] Ho HC, Mui M, Wan A, Ng YL, Stewart SM, Yew C, Lam TH, Chan SS. Happy Family Kitchen II: A Cluster Randomized Controlled Trial of a Community-Based Family Intervention for Enhancing Family Communication and Well-being in Hong Kong. Front Psychol. 2016 May 3;7:638. doi: 10.3389/fpsyg.2016.00638. eCollection 2016. PMID 27199864